CLINICAL TRIAL: NCT02122809
Title: Phase I Safety and Pharmacokinetics Study of Chiauranib in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Chiauranib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR101
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors
Keywords: Chiauranib, advanced solid tumors, phase 1 study
MeSH Terms: interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chiauranib (Experimental): Patients take a single dose of Chiauranib capsules for the pharmacokinetic study,then off for 5 days before the first cycle begins. In the subsequent treatment cycles, Chiauranib capsules are given orally once daily, 28 days as a cycle.
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — Take orally
  Other Names: CS2164

SUMMARY:
The purpose of this dose-escalation study is to assess the safety and tolerability of treatment with Chiauranib administered orally over a range of doses in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The purpose of this study is to assess the tolerability and safety include adverse events, vital signs, laboratory tests ,etc., of a range of doses of Chiauranib in solid tumor patients, and to determine the dose limit toxicity and the maximum tolerable dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of advanced solid tumor, including non-small cell lung cancer, colorectal cancer, ovarian cancer, renal cell carcinoma, gastrointestinal stromal tumor, gastric cancer, et al;
2. Patients with advanced solid tumors refractory to standard therapy or for which no standard therapy exists;
3. Body mass index (BMI) is between 18 and 28;
4. Age: 18~65 years;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
6. Laboratory criteria are as follows:

   1. Complete blood count: hemoglobin (Hb) ≥100g/L (no blood transfusion within 14 days); absolute neutrophil count (ANC) ≥1.5×109/L ; platelets >=100×109/L
   2. Biochemistry test: serum creatinine <=1.5×upper limit of normal (ULN); total bilirubin≦1.5×ULN; alanine aminotransferase / aspartate aminotransferase≦1.5×ULN; fasting triglyceride (TG) <= 3.0 mmol/L; total cholesterol <= 7.75 mmol/L
   3. Coagulation test: International Normalized Ratio (INR) < 1.5
7. Women of child-bearing potential should be non-lactating patients, and must agree to use effective contraceptive methods prior to study entry, during study participation, and up to 6 months following completion of therapy. A serum or urine pregnancy test within 7 days before enrollment must be negative; Men must agree to use effective contraceptive methods during study participation and up to 6 months following completion of therapy;
8. Willingness to sign a written informed consent document

Exclusion Criteria:

1. Life expectation < 3 months;
2. Subjects received anti-cancer therapy (including chemotherapy, radiotherapy, targeted therapy and endocrine therapy, et al) within 4 weeks prior to study entry; Subjects received nitrosoureas or mitomycin chemotherapy within 6 weeks prior to study entry;
3. Have uncontrolled or significant cardiovascular disease, including:

   1. Myocardial infarction (< the last 12 months)
   2. Uncontrolled angina (< the last 6 months)
   3. Congestive heart failure (< the last 6 months), or Left Ventricular Ejection Fraction (LVEF) < 50% prior to study entry
   4. History of any significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or TdP)
   5. History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 450 ms prior to study entry
   6. History of cerebrovascular accident
   7. Symptomatic coronary heart disease requiring treatment with agents
   8. Uncontrolled hypertension (> 140/90 mmHg) by single agent;
4. Have active bleeding , current thrombotic disease, or patients with bleeding potential receiving anticoagulation therapy;
5. History of deep vein thrombosis or pulmonary embolism;
6. Have unsolved toxicities (> grade 1) from prior anti-cancer therapy;
7. Have clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, that would impair the ingestion,transportation or absorption of oral agents, or patients undergone gastrectomy;
8. Have symptomatic brain metastasis;
9. History of organ transplantation;
10. Proteinuria positive;
11. Congenital or acquired immunodeficiency, active infections;
12. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document or the operation and compliance of study;
13. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | day 1-28
Number of Adverse Events | An expected average of 8 months

SECONDARY OUTCOMES:
pharmacokinetic profile of Chiauranib | On day 1,8,15,22,25,26,27,28
Evidence of benefit | An expected average of 8 months
  clinical benefit rate (complete response (CR),partial response (PR),stable disease (SD) > 8 weeks),duration of response (DOR),time to progression (TTP), or tumor marker improvement, if appropriate
Pharmacodynamic profile of Chiauranib | On day 15,28
  Plasma biomarkers: soluble vascular endothelial growth factor receptors (sVEGFR2), vascular endothelial growth factor (VEGF) Tumor tissue biomarkers: Aurora B, phospho-histone H3

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Yang L, Hao X, Liu Y, Zhang J, Ning Z, Shi Y. Phase I dose-escalation study of chiauranib, a novel angiogenic, mitotic, and chronic inflammation inhibitor, in patients with advanced solid tumors. J Hematol Oncol. 2019 Jan 14;12(1):9. doi: 10.1186/s13045-018-0695-0. PMID 30642372